CLINICAL TRIAL: NCT05159375
Title: The Effect of Protein Hydrolysate Supplementation to Influence the Expression of Strength Recovery and Systemic Muscle Function Markers Following Resistance Type Exercise in Male Subjects.
Brief Title: Effects of Protein Hydrolysate Supplementation Influencing Strength Recovery and Expression of Muscle Damage Markers Post-exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: Sports Surgery Clinic, Santry, Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PN20.004.01
Record Dates: First submitted 2021-09-27; First posted 2021-12-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-06

CONDITIONS: Muscle Injury
Keywords: muscle; function; markers; resistance; exercise; protein; hydrolysate; supplement; Elio
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elio (supplement under investigation) (Experimental): 2.4g of Elio administered orally daily with the first meal of the day for a 17 day period
  Interventions: Dietary Supplement: Elio
- Placebo (Placebo Comparator): 2.4g of SMCC administered orally daily with the first meal of the day for a 17 day period
  Interventions: Other: SMCC

INTERVENTIONS:
Dietary Supplement: Elio — Elio™ supplementation, a protein hydrolysate derived from fava bean protein extract
  Arms: Elio (supplement under investigation)
Other: SMCC — Placebo comparator
  Arms: Placebo

SUMMARY:
A randomised placebo controlled, double-blind, 30 Volunteer trial of Elio™ administered 2.4 grams per day in assessing its effects on post-exercise strength recovery and increases in markers associated with muscle injury and exertion.

DETAILED DESCRIPTION:
Periods of intense physical activity and exertion can lead to disruption of normal muscle homeostasis and the resultant muscle injury and recovery can impact upon quality of life especially in adult populations. Recovery post-exercise is therefore important to all active people.

There is a link between high-intensity exercise and reduced power and performance in the following exercise sessions. The effect on performance is measures as a reduced muscle force production or loss in strength and can correlate with delayed onset muscle soreness (DOMS). The reduced power/performance seen 24 hours - 7days post-exercise is affected by recovery methods applied, individual fitness levels and intensity of exercise injury.

Several theories have been proposed to explain the mechanisms underlying DOMS. These include inflammation and muscle damage.

Exercise-induced muscle damage is a transient phenomenon caused by unfamiliar, damaging exercise and is characterized by structural damage to myofibers and secondary inflammation. Signs and symptoms often persist for several days after exercise and typically include muscle soreness, elevated blood levels of intramuscular enzymes such as creatine kinase (CK), lactate dehydrogenase (LDH) and myoglobin (MB) that often result in elevations in circulating markers of inflammation such as C-reactive protein (CRP) and various interleukins. To date, extensive research has been published that explore the many recovery strategies purported to minimize indirect markers of muscle damage.

However, from a nutritional standpoint the results are weak. It is therefore important to develop nutritional products that can lessen the impact of these injuries' individuals succumb to or expedite their recovery.

Nutritional recovery strategies purported to minimise indirect markers of muscle damage and improve the inflammatory response can positively influence the recovery process after damaging exercise.

These strategies could in turn be used to prime the muscle for physical challenges.

Furthermore, there is a clear absence of natural approaches with proven evidence to address DOMS and the resulting performance declines.

Therapies such as non-steroidal anti-inflammatory drugs (NSAIDs) can be taken in the short term to reduce DOMS associated pain and inflammation. However, these drugs do not address performance strength loss linked to DOMS.

Acute injuries to discrete muscle groups can be indirectly detected by an array of systemic biomarkers, which become elevated at various time-points following the event.

This array of biomarkers represents key biochemical processes in muscle homeostasis, cellular integrity, mitochondrial function and inflammation.

Preliminary investigations in vitro and in vivo suggest that the administration of peptides isolated from the protein extract of fava beans, which constitute Elio™, can augment muscle protein synthesis (i.e. phospo-S6) and attenuate proteolytic signaling (i.e. Fbxo32 and Trim63) and surrogate inflammatory markers (TNFα and IL6). Thus, supporting the use of this hydrolysate in maintaining muscle homeostasis and function.

With the present study the investigators will investigate whether daily dietary supplementation of Elio™, over the course of 15 days can prime the muscle by improving strength recovery and attenuating the expression of systemic markers associated with muscle injury and over exertion following resistance type exercise in a healthy male population.

Objectives

To determine the effect of Elio™ supplementation, a protein hydrolysate derived from fava bean protein extract, on strength recovery and markers of muscle health, injury and function following strenuous resistance type exercise in male volunteers, aged between 30 and 45 years old following 17 days of supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Males between 30 and 45 years of age
2. Participants agree to comply with study procedures. Participants agree to comply with study procedures.
3. Participants agree to abstain from taking additional supplements throughout the testing period, with particular emphasis placed upon protein-based products
4. Participants agree to maintain their normal diet and exercise routine throughout the study
5. BMI between 18.5 to 29.9 kg/m2
6. Participants agree to refrain from consuming alcohol in the 48 hrs leading up to a test day.
7. Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits.
8. Provide voluntary, written, informed consent to participate in the study.
9. Refrain from any sort of exhaustive physical exercise from 48 hrs prior to each test or blood draw
10. Healthy as determined by medical examination at screening visit
11. Willingness to complete food diaries during the study
12. Must have a smart phone to use the Nutritics App
13. Non-smoker

Exclusion Criteria:

1. Alcohol or drug abuse in past year
2. Participation in any other clinical trial in the last 3 months from time of randomisation
3. Volunteer has a known allergy to the test material's active or inactive ingredients
4. Volunteers with unstable medical conditions
5. Any complaints that could interfere with ability to exercise
6. Individuals who are cognitively impaired and/or who are unable to give informed consent
7. Any co-morbidities interacting with mobility or muscle metabolism of the lower limbs (e.g., arthritis, spasticity/rigidity, all neurological disorders and paralysis)
8. Creatine supplements, anticoagulants, corticosteroids, growth hormones,

   testosterone, immunosuppressants, or exogenous insulin over the previous three months
9. Presence or history of neurological disorders or significant psychiatric illness.
10. Any other condition which in the Investigator's opinion may adversely affect the volunteer's ability to complete the study or its measures or which may pose significant risk to the volunteer
11. Participation in resistance or aerobic exercise within 48 hours of the test days
12. Participation in > 3 High-intensity Exercise sessions per Week
13. Undertake no recovery methods such as sea swims, foam rolling, cryotherapy or undue stretching during Days 14-17.
14. Have been in contact with a suspected or confirmed case of Covid-19 in the previous 14 days
15. Are Hepatitis A or B positive, HIV positive or have had a sexual partner who is infected with hepatitis or HIV

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in strength recovery | Two days
  Change in strength recovery post-resistance exercise as measured by peak torque from an isokinetic leg extension strength test between groups, ELIOTM and Placebo, at day 16 and day 17.

SECONDARY OUTCOMES:
Alteration in CK | Three days
  Attenuation of post-resistance exercise increases in creatine kinase (CK) as measured by ELISA compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker IL-6 | Three days
  Attenuation of post-resistance exercise alterations in IL-6 marker (pg/mL) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker LDH | Three days
  Attenuation of post-resistance exercise alterations in LDH marker (U/L) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker CRP | Three days
  Attenuation of post-resistance exercise alterations in CRP marker (μL/mL) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker MB | Three days
  Attenuation of post-resistance exercise alterations in MB marker (nM/L) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker TNF-α | Three days
  Attenuation of post-resistance exercise alterations in Tissue Necrosis Factor-α (TNFα) marker (pg/mL) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker Acylcarnitine | Three days
  Attenuation of post-resistance exercise alterations in Acylcarnitine marker (nMol/mL) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker FFA | Three days
  Attenuation of post-resistance exercise alterations in Free Fatty Acids (FFA) marker (mmol/L) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.
Alterations in muscle marker NAD+ | Three days
  Attenuation of post-resistance exercise alterations in NAD+ marker (arbitrary units) related to muscle homeostasis compared to Placebo after 14 days, 16 days and 17 days post-resistance exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Franklyn-Miller, Principal Investigator — Santry Sports Clinic
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Herrlinger KA, Chirouzes DM, Ceddia MA. Supplementation with a polyphenolic blend improves post-exercise strength recovery and muscle soreness. Food Nutr Res. 2015 Dec 18;59:30034. doi: 10.3402/fnr.v59.30034. eCollection 2015. PMID 26689317
- [Result] Clarkson PM, Hubal MJ. Exercise-induced muscle damage in humans. Am J Phys Med Rehabil. 2002 Nov;81(11 Suppl):S52-69. doi: 10.1097/00002060-200211001-00007. PMID 12409811
- [Result] Howatson G, van Someren KA. The prevention and treatment of exercise-induced muscle damage. Sports Med. 2008;38(6):483-503. doi: 10.2165/00007256-200838060-00004. PMID 18489195
- [Result] Cleak MJ, Eston RG. Delayed onset muscle soreness: mechanisms and management. J Sports Sci. 1992 Aug;10(4):325-41. doi: 10.1080/02640419208729932. PMID 1518094
- [Result] Ranchordas MK, Rogerson D, Soltani H, Costello JT. Antioxidants for preventing and reducing muscle soreness after exercise: a Cochrane systematic review. Br J Sports Med. 2020 Jan;54(2):74-78. doi: 10.1136/bjsports-2018-099599. Epub 2018 Jul 27. PMID 30054340